CLINICAL TRIAL: NCT00135005
Title: A Phase I Multicenter, Dose Escalation Study of AMN107 in Combination With Imatinib on a Continuous Daily Dosing Schedule in Adult Patients With Imatinib-resistant Gastrointestinal Stromal Tumors (GIST)
Brief Title: Study of AMN107 With Imatinib in Gastrointestinal Stromal Tumors (GIST)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107A2103; 2005-000561-18 (EudraCT Number)
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2013-05

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: GIST; AMN107; Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — nilotinib; Imatinib Mesylate

ARMS (1):
- AMN107 + STI571 (Experimental)
  Interventions: Drug: AMN107, STI571

INTERVENTIONS:
Drug: AMN107, STI571

SUMMARY:
This study is an open-label, multicenter, Phase I dose-escalation study of the combination of AMN107 and imatinib (STI571) in patients with imatinib-resistant GIST. This study is designed to determine the Phase II dose of AMN107 and imatinib when administered together in patients with imatinib-resistant GIST, and to characterize the safety, tolerability and pharmacokinetic (PK) profile of this combination.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastrointestinal stromal tumor (GIST).
* Patients who have had disease progression during imatinib therapy with 800 mg.
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with prior or concomitant malignancies other than GIST with the exception of previous or concomitant basal cell skin cancer or previous cervical carcinoma in situ.
* A history of impaired cardiac function or uncontrolled cardiovascular disease.
* Severe and/or uncontrolled concurrent disease that could cause unacceptable safety risks such as impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of AMN107.
* Currently taking certain medications that could affect an electrocardiogram result.
* Women who are pregnant or breast feeding.
* Patients unwilling or unable to comply with the protocol.

NOTE: Additional inclusion and/ or exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2005-08; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
To determine the MTD which will be the Phase II dose of AMN107 when given in combination with Imatinib. The MTD is defined to be the highest dose of AMN107 in combination with Imatinib given for at least 21 days in the first treatment cycle | From day 1 cycle 1 until at least six subjects have been treated at the recommended dose level and observed for at least 21 days
  MTD is defined to be the highest dose of AMN in combination with imatinib given for at least 21 days in the first treatment cycle

SECONDARY OUTCOMES:
To characterize safety and tolerability of AMN107 in combination with Imatinib in GIST | From day 1 cycle to the study completion visit
patients showing progression of disease on Imatinib. The patient will be followed-up for at least 4 cycles (28 days for one cycle) | up to 4 cycles after disease profression on imatinib
  cycle = 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (2):
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Philadelphia, Pennsylvania
- Novartis Investigative Site, Lyon, France
- Novartis Investigative Site, Berlin, Germany
- Novartis Investigative Site, Milan, MI, Italy

REFERENCES:
- See also: Results for CAMN107A2103 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=2942